CLINICAL TRIAL: NCT02696902
Title: A Phase 2 Proof-of-concept Study to Evaluate the Efficacy and Safety of MEDI3902 in Mechanically Ventilated Patients for the Prevention of Nosocomial Pneumonia Caused by Pseudomonas Aeruginosa
Brief Title: Effort to Prevent Nosocomial Pneumonia Caused by Pseudomonas Aeruginosa in Mechanically Ventilated Subjects
Acronym: EVADE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Collaborators: Innovative Medicines Initiative (Other); Antibacterial Resistance Leadership Group (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: D5470C00004
Record Dates: First submitted 2016-02-11; First posted 2016-03-02 (Estimated); Results first posted 2020-12-23 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-01

CONDITIONS: Pseudomonas Aeruginosa
Keywords: Pseudomonas aeruginosa, Pneumonia
MeSH Terms: conditions — Pseudomonas Infections; Pneumonia | interventions — gremubamab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- MEDI3902 500 mg (Experimental): Participants will receive a single intravenous (IV) dose of 500 mg MEDI3902.
  Interventions: Drug: MEDI3902
- Placebo (Placebo Comparator): Participants will receive a single IV dose of placebo matched to MEDI3902.
  Interventions: Other: Placebo
- MEDI3902 1500 mg (Experimental): Participants will receive a single IV dose of 1500 mg MEDI3902.
  Interventions: Drug: MEDI3902

INTERVENTIONS:
Drug: MEDI3902 — Participants will receive a single IV dose of MEDI3902 500 mg and 1500 mg in MEDI3902 500 mg arm and MEDI3902 1500 mg arm, respectively.
  Arms: MEDI3902 1500 mg; MEDI3902 500 mg
Other: Placebo — Participants will receive a single IV dose of placebo matched to MEDI3902.
  Arms: Placebo

SUMMARY:
Clinical trial looking to evaluate the efficacy and safety of MEDI3902 in mechanically ventilated participants for the prevention of nosocomial pneumonia caused by Pseudomonas aeruginosa.

ELIGIBILITY:
Inclusion Criteria:

Colonized with P aeruginosa, expected to require prolonged intubation and mechanical ventilation, without any evidence of active pneumonia.

Exclusion Criteria:

P aeruginosa disease at randomisation; lung injury score consistent with pneumonia; current lung disease; currently receiving protocol-specified Anti-P aeruginosa antibiotics, moribund participants.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2016-03-25 (Actual); Primary Completion 2019-12-04 (Actual); Study Completion 2019-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MedImmune LLC, Study Director — MedImmune LLC
Locations (66):
- United States (8):
  - Research Site, Englewood, Colorado
  - Research Site, Gainesville, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Augusta, Georgia
  - Research Site, Annapolis, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Cincinnati, Ohio
- Austria (2):
  - Research Site, Innsbruck
  - Research Site, Vienna
- Belgium (6):
  - Research Site, Bruges
  - Research Site, Brussels
  - Research Site, Genk
  - Research Site, Ghent
  - Research Site, Haine-Saint-Paul
  - Research Site, Ottignies
- Research Site, Slavonski Brod, Croatia
- Czechia (5):
  - Research Site, Brno
  - Research Site, Děčín
  - Research Site, Kolín
  - Research Site, Kyjov
  - Research Site, Teplice
- France (14):
  - Research Site, Argenteuil
  - Research Site, Clermont-Ferrand
  - Research Site, Garches
  - Research Site, La Tronche
  - Research Site, Le Kremlin-Bicêtre
  - Research Site, Le Plessis-Robinson
  - Research Site, Lille
  - Research Site, Limoges
  - Research Site, Montpellier
  - Research Site, Nancy
  - Research Site, Paris
  - Research Site, Pierre-Bénite
  - Research Site, Strasbourg
  - Research Site, Tours
- Greece (3):
  - Research Site, Athens
  - Research Site, Larissa
  - Research Site, Thessaloniki
- Hungary (3):
  - Research Site, Budapest
  - Research Site, Kistarcsa
  - Research Site, Vác
- Research Site, Dublin, Ireland
- Israel (4):
  - Research Site, Jerusalem
  - Research Site, Petah Tikva
  - Research Site, Ramat Gan
  - Research Site, Tel Aviv
- Portugal (3):
  - Research Site, Almada
  - Research Site, Lisbon
  - Research Site, Viana do Castelo
- Spain (11):
  - Research Site, Barcelona
  - Research Site, Córdoba
  - Research Site, Getafe
  - Research Site, Madrid
  - Research Site, Oviedo
  - Research Site, San Sebastián de los Reyes
  - Research Site, Santander
  - Research Site, Tarragona
  - Research Site, Terrassa
  - Research Site, Valencia
  - Research Site, Valladolid
- Turkey (Türkiye) (3):
  - Research Site, Ankara
  - Research Site, Istanbul
  - Research Site, Trabzon
- United Kingdom (2):
  - Research Site, Edgbaston
  - Research Site, London

REFERENCES:
- [Derived] Chastre J, Francois B, Bourgeois M, Komnos A, Ferrer R, Rahav G, De Schryver N, Lepape A, Koksal I, Luyt CE, Sanchez-Garcia M, Torres A, Eggimann P, Koulenti D, Holland TL, Ali O, Shoemaker K, Ren P, Sauser J, Ruzin A, Tabor DE, Akhgar A, Wu Y, Jiang Y, DiGiandomenico A, Colbert S, Vandamme D, Coenjaerts F, Malhotra-Kumar S, Timbermont L, Oliver A, Barraud O, Bellamy T, Bonten M, Goossens H, Reisner C, Esser MT, Jafri HS; COMBACTE-MAGNET EVADE Study Group. Safety, efficacy, and pharmacokinetics of gremubamab (MEDI3902), an anti-Pseudomonas aeruginosa bispecific human monoclonal antibody, in P. aeruginosa-colonised, mechanically ventilated intensive care unit patients: a randomised controlled trial. Crit Care. 2022 Nov 15;26(1):355. doi: 10.1186/s13054-022-04204-9. PMID 36380312
- See also: Redacted CSP for CT.gov results — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5470C00004&attachmentIdentifier=4b147617-87bc-4d06-bbb6-af4264ed0f66&fileName=CSP_EVADE_D5470C00004-Amendment_3_REDACTED_FINAL_01Dec20.pdf&versionIdentifier=
- See also: D5470C00004 Redacted SAP for CT.gov results — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5470C00004&attachmentIdentifier=0f441439-cf44-426d-8bde-f105d6c56781&fileName=D5470C00004_SAP_FINAL_v3.0_approved_REDACTED_FINAL_01Dec20.docx.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 188 participants were assigned to the study treatment groups. Out of 188 participants, 4 participants did not receive the study treatment.
Groups:
- Placebo: Participants received single intravenous (IV) dose of placebo matched to MEDI3902.
- MEDI3902 500 mg: Participants received single IV dose of 500 mg MEDI3902.
- MEDI3902 1500 mg: Participants received single IV dose of 1500 mg MEDI3902.
Period: Overall Study
Arm/Group | Placebo | MEDI3902 500 mg | MEDI3902 1500 mg
Started | 85 | 16 | 87
Treated | 83 | 16 | 85
Intent-to-treat (ITT) Population | 85 | 16 | 87
As-treated Population | 83 | 16 | 85
Modified Intent-to-treat (mITT) Population | 83 | 16 | 85
Completed | 63 | 12 | 59
Not Completed | 22 | 4 | 28
Not completed — Lost to Follow-up | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Death | 19 | 3 | 24
Not completed — Participant not fit post-randomization | 0 | 0 | 1
Not completed — Participant not eligible (negative PCR) | 0 | 0 | 1
Not completed — Principal investigator's decision | 1 | 0 | 0
Not completed — Sponsor's decision | 1 | 0 | 0
Not completed — Transferred to other hospital | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population is all randomized participants, grouped according to assigned treatment.
Groups:
- Placebo: Of the 85 participants, 83 participants received single intravenous (IV) dose of placebo matched to MEDI3902.
- MEDI3902 1500 mg: Of the 87 participants, 85 participants received single IV dose of 1500 mg MEDI3902.
- Total: Total of all reporting groups
Arm/Group | Placebo | MEDI3902 500 mg | MEDI3902 1500 mg | Total
Number analyzed (Participants) | 85 | 16 | 87 | 188
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.4 (13.0) | 62.7 (9.3) | 60.6 (15.1) | 62.5 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 6 | 32 | 60
  Male | 63 | 10 | 55 | 128
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 0 | 0 | 1
  Black or African American | 4 | 0 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  White | 77 | 16 | 83 | 176
  Other | 2 | 0 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Nosocomial Pneumonia Caused by Pseudomonas Aeruginosa
Description: Percentage of participants with nosocomial pneumonia caused by Pseudomonas aeruginosa is reported.
Time Frame: Day 1 through Day 22
Population: The modified intent to treat (mITT) population included all randomized and treated participants, grouped according to assigned treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | MEDI3902 500 mg | MEDI3902 1500 mg
Number analyzed (Participants) | 83 | 16 | 85
Percentage of participants | 18.1 | 12.5 | 22.4
Statistical Analysis 1: Comparison: Placebo vs MEDI3902 1500 mg; Test type: Superiority; p = 0.491, Poisson regression with robust variance; Relative risk reduction = -23.7, 80% CI 2-sided [-83.8 to 16.8]

2. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. The TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug.
Time Frame: Day 1 through Day 50
Population: The As-treated population is all treated participants, grouped according to actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI3902 500 mg | MEDI3902 1500 mg
Number analyzed (Participants) | 83 | 16 | 85
Participants | 81 | 15 | 84

3. Primary Outcome: Number of Participants With Treatment-emergent Serious Adverse Events (TESAEs)
Description: An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Day 1 through Day 50
Population: The As-treated population is all treated participants, grouped according to actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI3902 500 mg | MEDI3902 1500 mg
Number analyzed (Participants) | 83 | 16 | 85
Participants | 35 | 4 | 38

4. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events of Special Interest (TEAESI)
Description: An AESI is one of scientific and medical interest specific event for understanding of the study drug and may require close monitoring and rapid communication by the investigator to the sponsor. An AESI may be serious or non-serious.
Time Frame: Day 1 through Day 50
Population: The As-treated population is all treated participants, grouped according to actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI3902 500 mg | MEDI3902 1500 mg
Number analyzed (Participants) | 83 | 16 | 85
Participants | 1 | 0 | 2

5. Secondary Outcome: Maximum Observed Concentration (Cmax) of MEDI3902
Description: The Cmax of MEDI3902 is reported.
Time Frame: Day 1 (predose; 0 and 8 hours post dose), Day 2, Day 4, Day 8, Day 15, Day 22, Day 29, and Day 50
Population: The As-treated population is all treated participants, grouped according to actual treatment received. Number of Subjects Analyzed denotes the number of participants evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | MEDI3902 500 mg | MEDI3902 1500 mg
Number analyzed (Participants) | 16 | 84
mcg/mL | 87.6 (23.9) | 299 (94.1)

6. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to Infinity (AUC0-inf) of MEDI3902
Description: The AUC0-inf of MEDI3902 is reported.
Time Frame: Day 1 (predose; 0 and 8 hours post dose), Day 2, Day 4, Day 8, Day 15, Day 22, Day 29, and Day 50
Population: The As-treated population is all treated participants, grouped according to actual treatment received. Number of participants analyzed denotes the number of participants evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: day*mcg/mL
Arm/Group | MEDI3902 500 mg | MEDI3902 1500 mg
Number analyzed (Participants) | 16 | 81
day*mcg/mL | 440 (135) | 1510 (675)

7. Secondary Outcome: Clearance (CL) of MEDI3902
Description: The CL of MEDI3902 from body after intrevanous administration of single dose is reported.
Time Frame: Day 1 (predose; 0 and 8 hours post dose), Day 2, Day 4, Day 8, Day 15, Day 22, Day 29, and Day 50
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: L/day
Arm/Group | MEDI3902 500 mg | MEDI3902 1500 mg
Number analyzed (Participants) | 16 | 81
L/day | 1.31 (0.638) | 1.27 (0.86)

8. Secondary Outcome: Percentage of Participants Maintaining MEDI3902 Serum Levels Above the Target Level (1.7 µg/mL) Through 21 Days Post Dose
Description: Percentage of participants maintaining MEDI3902 serum levels above the target level (1.7 µg/mL) through 21 days post dose is reported.
Time Frame: Day 1 (predose; 0 and 8 hours post dose), Day 2, Day 4, Day 8, Day 15, and Day 22
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | MEDI3902 500 mg | MEDI3902 1500 mg
Number analyzed (Participants) | 16 | 84
Percentage of participants | 50 | 80.6

9. Secondary Outcome: Terminal Elimination Half-life (t1/2) of MEDI3902
Description: The t1/2 of MEDI3902 is reported.
Time Frame: Day 1 (predose; 0 and 8 hours post dose), Day 2, Day 4, Day 8, Day 15, Day 22, Day 29, and Day 50
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: day
Arm/Group | MEDI3902 500 mg | MEDI3902 1500 mg
Number analyzed (Participants) | 16 | 81
day | 6.56 (4.03) | 5.65 (2.69)

10. Secondary Outcome: Number of Participants With Positive Anti-drug Antibodies (ADA) to MEDI3902 Treatment
Description: Number of participants with positive ADA to MEDI3902 treatment is reported. Persistent positive is defined as positive at >= 2 post-baseline assessments or positive at last post-baseline assessment. Transient positive is defined as negative at last post-baseline assessment and positive at only one post-baseline assessment or at >= 2 post-baseline assessments.
Time Frame: Day 1 (predose), Day 15, Day 29, Day 50
Population: The As-treated population is all treated participants, grouped according to actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI3902 500 mg | MEDI3902 1500 mg
Number analyzed (Participants) | 83 | 16 | 85
Participants
  Positive at baseline and post-baseline | 3 | 2 | 1
  Persistent positive | 4 | 2 | 4
  Transient positive | 2 | 2 | 8

ADVERSE EVENTS:
Time Frame: Day 1 through Day 50
Arm/Group | Placebo | MEDI3902 500 mg | MEDI3902 1500 mg
All-Cause Mortality (participants affected / at risk) | 19/83 | 3/16 | 24/85
Serious Adverse Events (participants affected / at risk) | 35/83 | 4/16 | 38/85
Other Adverse Events (participants affected / at risk) | 79/83 | 15/16 | 82/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=83) | MEDI3902 500 mg (N=16) | MEDI3902 1500 mg (N=85)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 5 (5) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pulseless electrical activity (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Deafness (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 1 (1) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 3 (3) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Acinetobacter bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Biliary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Brain abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Burkholderia cepacia complex infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Candida sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Endocarditis enterococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Escherichia sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Klebsiella bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Klebsiella sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia pseudomonal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pseudomonal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pseudomonal sepsis (Infections and infestations) | 4 (4) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 3 (3) | 0 (0) | 3 (3)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Weaning failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Oxygen saturation decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Brain injury (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Coma (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Device occlusion (Product Issues) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Polyuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 4 (4)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mediastinal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (4)
Shock (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=83) | MEDI3902 500 mg (N=16) | MEDI3902 1500 mg (N=85)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Anaemia of chronic disease (Blood and lymphatic system disorders) | 4 (5) | 0 (0) | 4 (4)
Blood loss anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Haemolytic anaemia (Blood and lymphatic system disorders) | 5 (9) | 0 (0) | 8 (13)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 7 (10) | 1 (1) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (2)
Microcytic anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0)
Normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Splenomegaly (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 4 (4)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 2 (2) | 4 (7)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 2 (2) | 0 (0) | 3 (5)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cyanosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Mitral valve stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 7 (11) | 0 (0) | 3 (3)
Ventricular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Excessive cerumen production (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetes insipidus (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Euthyroid sick syndrome (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperprolactinaemia (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1)
Blindness unilateral (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Noninfective conjunctivitis (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Pupils unequal (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 6 (6) | 2 (3) | 3 (6)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Aerophagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 11 (13) | 4 (5) | 11 (11)
Diarrhoea (Gastrointestinal disorders) | 11 (16) | 4 (5) | 12 (14)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 6 (6)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal hypomotility (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal oedema (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal dilatation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lip haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 3 (3) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (5) | 4 (5) | 1 (2)
Oesophagopleural fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oral mucosa haematoma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatic failure (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatic necrosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Perianal erythema (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Salivary hypersecretion (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (5) | 2 (4) | 4 (6)
Asthenia (General disorders) | 2 (2) | 0 (0) | 1 (1)
Catheter site inflammation (General disorders) | 2 (3) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0)
Complication associated with device (General disorders) | 0 (0) | 0 (0) | 2 (2)
Generalised oedema (General disorders) | 2 (2) | 0 (0) | 0 (0)
Granuloma (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperthermia (General disorders) | 2 (4) | 1 (1) | 2 (2)
Hypothermia (General disorders) | 2 (3) | 0 (0) | 2 (3)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Medical device pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Medical device site dermatitis (General disorders) | 0 (0) | 0 (0) | 1 (1)
Medical device site haemorrhage (General disorders) | 1 (2) | 0 (0) | 0 (0)
Mucosal ulceration (General disorders) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 4 (4) | 1 (1) | 3 (4)
Pain (General disorders) | 8 (15) | 0 (0) | 7 (7)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 13 (20) | 1 (1) | 16 (20)
Swelling (General disorders) | 1 (1) | 0 (0) | 0 (0)
Thirst (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatocellular injury (Hepatobiliary disorders) | 2 (2) | 0 (0) | 2 (2)
Ischaemic hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Acinetobacter infection (Infections and infestations) | 2 (2) | 0 (0) | 5 (5)
Anal fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 4 (4) | 0 (0) | 4 (5)
Bacterial abdominal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bacterial disease carrier (Infections and infestations) | 1 (2) | 0 (0) | 3 (5)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Bacterial sepsis (Infections and infestations) | 0 (0) | 0 (0) | 4 (4)
Bacteriuria (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchitis bacterial (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Candida infection (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Candiduria (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Citrobacter bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (3)
Conjunctivitis (Infections and infestations) | 1 (3) | 1 (1) | 0 (0)
Cystitis klebsiella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Empyema (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Enterobacter bacteraemia (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Enterobacter pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Enterococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Enterococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (2)
Enterococcal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 5 (5) | 1 (2) | 3 (4)
Eye infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fungaemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Genital infection female (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Haematoma infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Herpes virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Klebsiella bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 3 (3)
Klebsiella infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Klebsiella sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lung infection pseudomonal (Infections and infestations) | 2 (5) | 0 (0) | 1 (1)
Morganella infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 3 (3)
Oral fungal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 3 (3)
Pneumonia acinetobacter (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 12 (13) | 2 (2) | 4 (5)
Pneumonia escherichia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia proteus (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia pseudomonal (Infections and infestations) | 12 (13) | 1 (1) | 13 (15)
Pneumonia staphylococcal (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Proteus infection (Infections and infestations) | 4 (4) | 1 (2) | 1 (1)
Pseudomonal bacteraemia (Infections and infestations) | 6 (6) | 0 (0) | 6 (6)
Pseudomonal sepsis (Infections and infestations) | 5 (6) | 0 (0) | 0 (0)
Pseudomonas bronchitis (Infections and infestations) | 5 (5) | 4 (4) | 4 (4)
Pseudomonas infection (Infections and infestations) | 4 (4) | 0 (0) | 4 (4)
Pyuria (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Serratia bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Serratia sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 2 (2) | 1 (1) | 4 (4)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Stenotrophomonas infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Stoma site infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Systemic candida (Infections and infestations) | 3 (3) | 0 (0) | 1 (1)
Tracheobronchitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (2) | 3 (3)
Urinary tract infection bacterial (Infections and infestations) | 3 (3) | 0 (0) | 3 (3)
Urinary tract infection pseudomonal (Infections and infestations) | 5 (6) | 0 (0) | 4 (4)
Urinary tract infection staphylococcal (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Varicella zoster virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Dialysis related complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Eschar (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0)
Flail chest (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Gastrostomy tube site complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Haemodilution (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Inflammation of wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Palate injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Post procedural inflammation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Postoperative hypotension (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Procedural hypotension (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 3 (3)
Scar (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1)
Scratch (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Stoma site erythema (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Tracheal haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2)
Weaning failure (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 2 (2)
Wound necrosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Wound secretion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 4 (4) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 0 (0) | 0 (0)
Blood albumin decreased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Blood magnesium decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood potassium decreased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Blood sodium decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 3 (3)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Electrocardiogram qt prolonged (Investigations) | 0 (0) | 1 (1) | 1 (1)
Inflammatory marker increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Oxygen saturation abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Oxygen saturation decreased (Investigations) | 3 (9) | 0 (0) | 3 (10)
Pco2 increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Po2 decreased (Investigations) | 1 (3) | 0 (0) | 1 (5)
Transaminases increased (Investigations) | 1 (1) | 1 (1) | 1 (1)
Urine output decreased (Investigations) | 2 (2) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (3)
Alkalosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (6)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hyperammonaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 4 (5)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 3 (4)
Hypernatraemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 5 (5)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0) | 3 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 9 (12) | 1 (1) | 15 (25)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (4)
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2)
Metabolic alkalosis (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 4 (5)
Vitamin k deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Bone disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Exposed bone in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (3)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 3 (3) | 2 (2)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 3 (3)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Complex regional pain syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Frontotemporal dementia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (3) | 0 (0) | 4 (7)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Motor dysfunction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Myoclonus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Paresis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Parkinsonism (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Peripheral sensorimotor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Peroneal nerve palsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Post cardiac arrest syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Psychomotor hyperactivity (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Stent malfunction (Product Issues) | 1 (1) | 0 (0) | 0 (0)
Thrombosis in device (Product Issues) | 1 (1) | 0 (0) | 0 (0)
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 3 (3) | 1 (1) | 3 (3)
Anxiety (Psychiatric disorders) | 4 (5) | 3 (3) | 2 (2)
Apathy (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Compulsive lip biting (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 5 (5)
Depression (Psychiatric disorders) | 2 (2) | 0 (0) | 3 (3)
Depressive symptom (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Disinhibition (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Disorientation (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1)
Initial insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 9 (10) | 0 (0) | 7 (7)
Intensive care unit delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Nervousness (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 0 (0) | 1 (1)
Anuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 2 (2)
Haemorrhage urinary tract (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Oliguria (Renal and urinary disorders) | 5 (6) | 1 (1) | 5 (5)
Polyuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal cyst (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 3 (3) | 0 (0) | 5 (5)
Renal impairment (Renal and urinary disorders) | 1 (1) | 1 (1) | 2 (2)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Urinary tract disorder (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Urine abnormality (Renal and urinary disorders) | 1 (1) | 0 (0) | 2 (2)
Vesical fistula (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Cervical cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Genital pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Oedema genital (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Penile discharge (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Penile oedema (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus genital (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Vulval disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (1) | 4 (4)
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0)
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (2)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 5 (8)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Hypopnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 2 (2)
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Increased viscosity of bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 2 (2)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Pleural disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 3 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Pulmonary fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (5)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory fatigue (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sputum retention (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) | 3 (3)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 6 (6) | 0 (0) | 5 (6)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 3 (5) | 0 (0) | 2 (2)
Generalised erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 3 (5)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Scab (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin ulcer haemorrhage (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Artery dissection (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Extremity necrosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Haemodynamic instability (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 7 (9) | 3 (5) | 3 (6)
Hypoperfusion (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 16 (21) | 1 (1) | 23 (29)
Jugular vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral coldness (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Subclavian vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Vein disorder (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Venous thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.

DOCUMENTS (2):
  • Study Protocol (2018-06-06): https://cdn.clinicaltrials.gov/large-docs/02/NCT02696902/Prot_002.pdf
  • Statistical Analysis Plan (2020-02-17): https://cdn.clinicaltrials.gov/large-docs/02/NCT02696902/SAP_003.pdf